CLINICAL TRIAL: NCT06780111
Title: A Phase 1/2 Open-Label, Umbrella Platform Design Study of Investigational Agents in Combination With Pembrolizumab (MK-3475) With or Without Chemotherapy in Participants With 1L Locally Advanced Unresectable/Metastatic Esophageal Cancer: KEYMAKER-U06 Substudy 06E
Brief Title: Substudy 06E: Umbrella Study of Combination Therapies in Esophageal Cancer (MK-3475-06E/KEYMAKER-U06)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-06E; MK-3475-06E (Other: MSD); 2024-514273-22-00 (Registry Identifier: EU CT); U1111-1307-6484 (Registry Identifier: UTN); jRCT2041240166 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — pembrolizumab; Leucovorin; Levoleucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Pembrolizumab + Chemotherapy (Active Comparator): Participants will receive 400 mg of pembrolizumab via intravenous (IV) infusion every six weeks (Q6W) on Day 1 of each 42 day cycle up to 18 cycles (up to approximately 2 years), and mFOLFOX6 chemotherapy: oxaliplatin 85 mg/m^2 via IV infusion every 2 weeks (Q2W) until progressive disease (PD) or toxicity; leucovorin 400 mg/m2 OR levoleucovorin 200 mg/m^2 via IV infusion Q2W until PD or toxicity; 5-fluorouracil (5-FU) 400 mg/m^2 bolus IV infusion followed by 2400 mg/m^2 continuous 46-48 hour IV infusion Q2W until PD or toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Leucovorin; Drug: Levoleucovorin; Drug: 5-Fluorouracil (5-FU); Drug: Oxaliplatin
- Pembrolizumab + I-DXd (Experimental): Participants will receive 200 mg of pembrolizumab via IV infusion Q3W on Day 1 of each 21 day cycle for up to 35 cycles (up to approximately 2 years). Participants will also receive up to 12 mg/kg I-XDd Q3W via IV infusion until PD or toxicity.
  Interventions: Biological: Pembrolizumab; Biological: I-DXd; Drug: Rescue Medication
- Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin (Experimental): Participants will receive 200 mg pembrolizumab via IV infusion Q3W on Day 1 of each 21 day cycle up to 35 cycles (up to approximately 2 years). Participants will also receive I-DXd up to 12 mg/kg via IV infusion Q3W until PD or toxicity, 5-FU 400 mg/m^2 bolus IV infusion followed by 2400 mg/m^2 continuous 46-48 hour IV infusion Q2W until PD or toxicity, and leucovorin 400 mg/m^2 OR levoleucovorin 200 mg/m^2 via IV infusion Q2W until PD or toxicity.
  Interventions: Biological: Pembrolizumab; Biological: I-DXd; Drug: Leucovorin; Drug: Levoleucovorin; Drug: 5-Fluorouracil (5-FU); Drug: Rescue Medication
- Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin + Oxaliplatin (Experimental): Participants will receive 200 mg of pembrolizumab via IV infusion Q3W on Day 1 of each 21 day cycle up to 35 cycles (up to approximately 2 years). Participants will also receive up to 12 mg/kg I-DXd via IV infusion q3w until PD or toxicity, 5-FU 2400 mg/m^2 continuous 46-48 hour IV infusion Q2W until PD or toxicity, 60mg/m^2 oxaliplatin via IV infusion Q2W until PD or toxicity, and leucovorin 400 mg/m^2 OR levoleucovorin 200 mg/m^2 via IV infusion Q2W until PD or toxicity.
  Interventions: Biological: Pembrolizumab; Biological: I-DXd; Drug: Leucovorin; Drug: Levoleucovorin; Drug: 5-Fluorouracil (5-FU); Drug: Oxaliplatin; Drug: Rescue Medication
- Pembrolizumab + Sacituzumab tirumotecan + 5-FU IV + Leucovorin or Levoleucovorin (Experimental): Participants will receive 400 mg pembrolizumab via IV infusion Q6W on Day 1 of each 42 day cycle up to 18 cycles (up to approximately 2 years). Participants will also receive sacituzumab tirumotecan 4 mg/kg via IV infusion Days 1, 15, and 29 every 42 day cycle until PD or toxicity, 5-FU 400 mg/m^2 bolus IV infusion followed by 2400 mg/m^2 continuous 46-48 hour IV infusion Q2W until PD or toxicity, and leucovorin 400 mg/m^2 OR levoleucovorin 200 mg/m^2 via IV infusion Q2W until PD or toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Leucovorin; Drug: Levoleucovorin; Drug: 5-Fluorouracil (5-FU); Biological: Sacituzumab tirumotecan; Drug: Rescue Medication

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
Biological: I-DXd — IV infusion
  Other Names: Ifinatamab deruxtecan; MK-2400; DS-7300a
  Arms: Pembrolizumab + I-DXd; Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin; Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin + Oxaliplatin
Drug: Leucovorin — IV infusion
  Arms: Pembrolizumab + Chemotherapy; Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin; Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin + Oxaliplatin; Pembrolizumab + Sacituzumab tirumotecan + 5-FU IV + Leucovorin or Levoleucovorin
Drug: Levoleucovorin — IV infusion
  Arms: Pembrolizumab + Chemotherapy; Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin; Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin + Oxaliplatin; Pembrolizumab + Sacituzumab tirumotecan + 5-FU IV + Leucovorin or Levoleucovorin
Drug: 5-Fluorouracil (5-FU) — IV Infusion
  Arms: Pembrolizumab + Chemotherapy; Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin; Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin + Oxaliplatin; Pembrolizumab + Sacituzumab tirumotecan + 5-FU IV + Leucovorin or Levoleucovorin
Drug: Oxaliplatin — IV infusion
  Arms: Pembrolizumab + Chemotherapy; Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin + Oxaliplatin
Biological: Sacituzumab tirumotecan — IV infusion
  Other Names: MK-2870; SKB264
  Arms: Pembrolizumab + Sacituzumab tirumotecan + 5-FU IV + Leucovorin or Levoleucovorin
Drug: Rescue Medication — Includes 5-HT3 receptor antagonist, NK-1 receptor antagonist, and corticosteroid for Arms 2, 3, and 4, and H1 receptor antagonist, H2 receptor antagonist, acetaminophen, and dexamethasone for Arm 5, administered per approved product label
  Arms: Pembrolizumab + I-DXd; Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin; Pembrolizumab + I-DXd + 5-FU IV + Leucovorin or Levoleucovorin + Oxaliplatin; Pembrolizumab + Sacituzumab tirumotecan + 5-FU IV + Leucovorin or Levoleucovorin

SUMMARY:
Researchers are looking for new ways to treat esophageal squamous cell carcinoma (ESCC). ESCC is a type of cancer that starts in certain cells that line the esophagus. The esophagus is the tube that connects the throat to the stomach. This study will look at ESCC that is either locally advanced unresectable, which means it has spread into tissue near where it started and cannot be completely removed by surgery, or metastatic, which means it has spread to other body parts.

Available treatments for these types of ESCC include pembrolizumab and chemotherapy. Pembrolizumab is an immunotherapy, which is a treatment that helps the immune system fight cancer. Chemotherapy is medicine that destroys cancer cells or stops them from growing.

Researchers want to learn about giving pembrolizumab and investigational agents, with or without chemotherapy to treat ESCC. Ifinatamab deruxtecan (I-DXd), is an antibody-drug conjugate (ADC). An ADC attaches to a protein on cancer cells and delivers treatment to destroy those cells.

The main goal of this study is to learn about the safety of investigational agents and pembrolizumab with or without chemotherapy and if people tolerate them. Researchers also want to learn how cancer responds (gets smaller or goes away) to the study treatments.

DETAILED DESCRIPTION:
The master protocol is MK-3475-U06

ELIGIBILITY:
Inclusion Criteria

The main inclusion criteria include but are not limited to the following:

* Has histologically or cytologically confirmed diagnosis of locally advanced unresectable or metastatic squamous cell carcinoma of the esophagus in first-line (1L) setting.
* Has measurable disease per RECIST 1.1 as assessed by the local site. investigator or designee/radiology assessment and verified by BICR. Lesions situated in a previously irradiated area are considered measurable if progression has been shown in such lesions.
* Has AEs due to previous anticancer therapies of ≤Grade 1 or baseline (except alopecia and vitiligo). Endocrine-related AEs adequately treated with hormone replacement are acceptable.
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART).
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Has adequate organ function.

Exclusion Criteria

The main exclusion criteria include but are not limited to the following:

* Has had systemic anticancer therapy for locally advanced unresectable or metastatic esophageal cancer.
* Has tumor invasion into organs located adjacent to the esophageal disease site (eg, aorta or respiratory tract) at an increased risk of fistula.
* Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage or medical intervention.
* Has clinically significant corneal disease, history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Has received prior therapy with an anti-programmed cell death 1 protein (PD-1), anti-programmed cell death ligand 1 (PD-L1), or anti-programmed cell death ligand 2 (PD-L2) agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor.
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study intervention.
* Has received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Has inadequate cardiac function assessed as: - corrected QT interval by Fredericia (QTcF) value >470 msec.
* Has clinically significant cardiovascular disease within 6 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.
* Has peripheral neuropathy ≥ Grade 2.
* Has diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention.
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Has had (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease, and/or suspected interstitial lung disease (ILD)/pneumonitis that cannot be ruled out by imaging at Screening.
* Has active infection requiring systemic therapy.
* Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses, including, but not limited to, any underlying pulmonary disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2032-01-04 (Estimated); Study Completion 2032-01-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Experience Dose Limiting Toxicities (DLTs) During the Safety Lead-In Phase | Up to approximately 28 days
  Percentage of participants experiencing toxicities that are possibly, probably, or definitely related to study intervention; that meet pre-defined severity criteria; and result in a change in the given dose.
Percentage of Participants who Experience an Adverse Event (AE) | Up to approximately 77 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience an AE will be reported.
Objective Response Rate (ORR) | Up to approximately 77 months
  ORR is defined as a confirmed complete response (CR: the disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 as assessed by blinded independent central review (BICR). The percentage of participants who experience CR or PR as assessed by BICR will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 77 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression-Free Survival (PFS) | Up to approximately 77 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 77 months
  OS is defined as the time from allocation/randomization to death due to any cause.
Disease Control Rate (DCR) | Up to approximately 77 months
  DCR is defined as a confirmed complete response (CR) or partial response (PR), or stable disease (SD) with at least 6 months PFS per RECIST 1.1 as assessed by BICR.
Maximum Plasma Concentration (Cmax) of I-DXd | At designated time points up to approximately 65 months
  Cmax is defined as the peak level I-DXd reaches in the blood plasma. Blood samples collected predose and at multiple timepoints postdose will be used to determine the Cmax of I-DXd when co-administered with other investigational agents.
Time to Maximum Plasma Concentration (Tmax) of I-DXd | At designated time points up to approximately 65 months
  Tmax is defined as the time it took I-DXd to reach its peak level in blood plasma. Blood samples collected predose and at designated timepoints postdose will be used to determine the Tmax of I-DXd when co-administered with other investigational agents.
Area Under the Concentration-Time Curve from Time 0 to Last Measurable Plasma Concentration (AUClast) of I-DXd | At designated time points up to approximately 65 months
  AUClast is defined as the area under the concentration-time curve from time 0 to the last measurable concentration of I-DXd in the blood plasma. Blood samples collected at predose and at designated timepoints postdose will be used to determine the AUClast of I-DXd in combination with other agents.
Area Under the Concentration-Time Curve from Time 0 to the End of the Dosing Period (AUCtau) of I-DXd | At designated time points up to approximately 65 months
  AUCtau is defined as the area under the concentration-time curve from time zero to the end of the dosing period. Blood samples collected at predose and at designated timepoints postdose will be used to determine the AUCtau of I-DXd in combination with other agents.
The Percentage of Participants with Antidrug Antibodies (ADA) Against I-DXd | Up to approximately 65 months
  Blood samples collected at designated timepoints will be used to determine the ADA response to I-DXd. The percentage of participants with ADA will be reported.
The Percentage of Participants with Treatment-Emergent ADA Against I-DXd | Up to approximately 65 months
  Blood samples collected at designated timepoints will be used to determine the treatment-emergent ADA response to I-DXd. The percentage of participants who have treatment-emergent I-DXd ADA will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (41):
- UPMC Hillman Cancer Center ( Site 1904), Pittsburgh, Pennsylvania, United States
- Brazil (2):
  - Liga Norte Riograndense Contra o Cancer ( Site 1301), Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceicao ( Site 1300), Porto Alegre, Rio Grande do Sul
- Chile (6):
  - Clínica Puerto Montt ( Site 1406), Port Montt, Los Lagos Region
  - FALP ( Site 1400), Santiago, Region M. de Santiago
  - Centro de Oncología de Precisión ( Site 1402), Santiago, Region M. de Santiago
  - Clínica UC San Carlos de Apoquindo ( Site 1403), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 1401), Santiago, Region M. de Santiago
  - Bradford Hill Norte ( Site 1405), Antofagasta
- China (6):
  - The Second Affiliated Hospital of Anhui Medical University ( Site 9511), Hefei, Anhui
  - Beijing Cancer Hospital ( Site 9500), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University ( Site 9503), Xiamen, Fujian
  - Henan Cancer Hospital ( Site 9509), Zhengzhou, Henan
  - Xuzhou Central Hospital ( Site 9512), Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 9505), Nanchang, Jiangxi
- Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 9000), Brno, Brno-mesto, Czechia
- France (3):
  - C.H.R.U. de Brest - Hopital Cavale Blanche ( Site 9104), Brest, Finistere
  - CHU Lille - Institut Coeur Poumon ( Site 9100), Lille, Nord
  - Pitie Salpetriere University Hospital ( Site 9102), Paris
- Haematologisch-Onkologische Praxis Eppendorf Facharztzentrum Eppendorf - Hope ( Site 1807), Hamburg, Germany
- Italy (2):
  - Ospedale San Raffaele-Oncologia Medica ( Site 9201), Milan, Lombardy
  - Istituto Oncologico Veneto IRCCS ( Site 9202), Padua, Veneto
- Japan (3):
  - Aichi Cancer Center ( Site 9702), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 9701), Kashiwa, Chiba
  - National Cancer Center Hospital ( Site 9700), Chūō, Tokyo
- Oslo Universitetssykehus Radiumhospitalet ( Site 1501), Oslo, Norway
- National University Hospital ( Site 9800), Singapore, Central Singapore, Singapore
- South Korea (3):
  - National Cancer Center ( Site 9902), Goyang-si, Kyonggi-do
  - Asan Medical Center ( Site 9901), Seoul
  - Samsung Medical Center ( Site 9900), Seoul
- Switzerland (2):
  - Kantonsspital Graubuenden ( Site 1700), Chur, Kanton Graubünden
  - Hopitaux Universitaires de Geneve HUG. ( Site 1701), Geneva
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 1009), Kaoshiung, Kaohsiung
  - Kaohsiung Chang Gung Memorial Hospital ( Site 1003), Kaohsiung City
  - China Medical University Hospital ( Site 1007), Taichung
  - National Cheng Kung University Hospital ( Site 1001), Tainan
  - National Taiwan University Hospital ( Site 1000), Taipei
  - Taipei Veterans General Hospital ( Site 1005), Taipei
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 1006), Taoyuan District
- Thailand (2):
  - Ramathibodi Hospital ( Site 1103), Ratchathewi, Bangkok
  - Songklanagarind hospital ( Site 1101), Hat Yai, Changwat Songkhla

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com